CLINICAL TRIAL: NCT04627077
Title: Livestrong Cancer Institutes' Patient Reported Outcomes Study
Acronym: LCI PROs
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Gail Eckhardt, Director, LIVESTRONG Cancer Institutes Chair, Department of Oncology, University of Texas at Austin
Other Study IDs: 2017-08-0081
Record Dates: First submitted 2018-05-04; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Neoplasms; Drug Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SIC drug therapy patients: Patients with a cancer diagnosis currently being treated at SIC clinic

SUMMARY:
The goal of this study will be to collect baseline patient reported outcome measures at the Livestrong Cancer Institutes (LCI) with the goal of improving quality care and to inform decision making by patients, providers, and researchers for future LCI initiatives.

DETAILED DESCRIPTION:
This proposed study is a descriptive study of the adult oncology population at the Seton Infusion Center in order to provide information about patient needs and identify areas for further research and resource allocation. The patient reported outcome measures being collected cover the following domains: anxiety, depression, fatigue, physical function, financial toxicity and pain. Patients and caregivers will be informed about the study and given the opportunity to enroll at the time of routine clinic visits at the Dell Seton Medical Center at The University of Texas Seton Infusion Center (SIC). Patients choosing to enroll in the study will be provided informed consent, and then allowed to complete the measures during their clinic visit on an iPad provided by the research staff. After IRB approval for a period of 1-2 months data collection will take place at the SIC clinic at DMS. Upon completion of the measures patients will be asked for an email address and phone number so that a follow up link to survey questions can be sent to them in 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and older, being treated for cancer at the Seton Infusion Clinic
* Patient cognitively and physically able to complete questionnaires on an ipad in English or Spanish.

Exclusion Criteria:

* -Patient unable to speak English or Spanish as required for study data collection
* Patient cognitively or physically unable to complete measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total sample size of 200 adult patients and caregivers (n=200 dyads). Patients are currently receiving treatment for a cancer diagnosis at the Seton Infusion Center.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life - FACT-G | Baseline
  Functional Assessment of Cancer Therapy (FACT-G)
Change in Anxiety - PROMIS | Baseline and 3 month follow up
  PROMIS adaptive anxiety
Change in Depression - PROMIS | Baseline and 3 month follow up
  PROMIS adaptive Depression
Change in Pain - PROMIS | Baseline and 3 month follow up
  PROMIS adaptive pain
Change in Physical Function- PROMIS | Baseline and 3 month follow up
  PROMIS adaptive physical function
Change in Fatigue - PROMIS | Baseline and 3 month follow up
  PROMIS adaptive fatigue
Change in Financial Toxicity | Baseline and 3 month follow up
  Comprehensive Score for financial Toxicity (COST) questionnaire
Change in Patient satisfaction with care | Baseline and 3 month follow up
  The CAHPS® Cancer Care Survey

SECONDARY OUTCOMES:
Change in Impact on Caregivers | Baseline and 3 month follow up
  Brief Assessment Scale for Caregivers (BASC), range -27 to 12, higher scores poorer outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Seton Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No